CLINICAL TRIAL: NCT00001471
Title: Virologic and Immunologic Evaluation of Lymph Node, Tonsillar and Intestinal Biopsies, and Bronchoalveolar Lavage Fluid
Brief Title: Tissue Biopsy and Imaging Studies in HIV-Infected Patients
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950027; 95-I-0027
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-09-10

CONDITIONS: HIV; ICL; Healthy Volunteers
Keywords: AIDS; HIV; Retrovirus; Therapy; Response; Natural History
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Healthy Volunteers
- HIV-infected: HIV-infected individuals
- ICL: Idiopathic CD4 lymphopenia

SUMMARY:
This study will examine tissue from the tonsils, lymph nodes and large bowel of HIV-infected patients to investigate changes in viral load and certain white blood cells during treatment.

Normal volunteers and HIV-infected patients 18 years of age or older may be eligible for this study. Candidates will be screened with a medical history, physical examination, blood and urine tests and possibly an electrocardiogram (EKG). Blood tests may include HLA typing, a genetic test of immune system markers.

Participants may undergo the following procedures:

* Blood tests (patients and volunteers)
* Biopsies The frequency of biopsies for given patients may vary, depending on their specific therapy. Typically, biopsies are done at a single time, or for patients starting a new therapy, biopsies could be performed before starting therapy, during therapy and possibly after completion of therapy.
* Tonsil biopsies (patients and volunteers) Volunteers will have one tonsil biopsy. Patients will have no more than six tonsil biopsies, with no more than three in a 10-day period. The biopsy is done by an ear, nose and throat specialist as an outpatient procedure. The tonsils are numbed with a local anesthetic, and one to four pieces of tissue are extracted.
* Lymph node biopsies (patients only) Patients will have no more than four lymph node biopsies, performed no more frequently than once a month. The biopsy is done by a surgeon and may require a 2- to 3-day hospital stay. The skin above the lymph nodes is numbed with a local anesthetic, an incision is made and the tissue is removed. Alternatively, a needle biopsy may be done, in which a small amount of lymph tissue is withdrawn through a special needle injected into the site.
* Intestinal biopsies (patients and volunteers) Volunteers will have one intestinal biopsy procedure. Patients may have up to six intestinal biopsy procedures, each separated by at least 10 days. This is done by a gastroenterologist as an outpatient procedure. A flexible tube (sigmoidoscope or colonoscope) with a light and special lens at the tip is inserted into the rectum and large bowel. Wire instruments passed through the tube are used to extract small tissue samples.
* Bronchoalveolar lavage (BAL; patients and volunteers) Volunteers and patients will undergo bronchoscopy in which a flexible tube (bronchoscope) with a light and special lens at the tip is inserted through the nose or mouth into the lungs, and the lining of the lung is sampled by washing the airways with small amounts of saline. The procedure is performed by a pulmonologist or critical care specialist, usually as an outpatient.

DETAILED DESCRIPTION:
Examining tissues outside the bloodstream in HIV-infected patients, patients with Idiopathic CD4 lymphopenia (ICL) and, for comparison, HIV-uninfected healthy volunteers (hereafter referred to as healthy volunteers), can provide insights into the pathogenesis of HIV infection and ICL. This protocol will provide a mechanism for sampling tissue sites. A total of 430 HIV-infected patients, 100 ICL patients and 105 healthy volunteers will be enrolled in these studies. To assess changes in viral load and immunological parameters at sites outside the bloodstream during therapy of HIV-infected patients, sequential tonsillar, lymph node, or intestinal biopsies, or bronchoscopy with bronchoalveolar lavage (BAL) will be undertaken during the course of therapy. In a small number of patients, sequential or simultaneous lymph node biopsies will be performed. In addition, uninfected healthy volunteers will be enrolled to have a tonsillar or intestinal biopsy, or bronchoscopy with BAL; this will allow comparison of immunologic parameters in HIVinfected and uninfected tonsillar or intestinal tissues, or BAL fluid. Finally, ICL patients may have tissue sampling to assess lymphocyte distribution and possible function in tissues to better understand the pathogenesis of their lymphopenia. Sequential or simultaneous tissue sampling may occur and longitudinal samples may also be obtained to assess stability in tissue compartments or effect of possible immunomodulatory treatments.

ELIGIBILITY:
* INCLUSION CRITERIA:

Greater than or equal to 18 years old.

Ability to sign informed consent.

For women of child-bearing potential, negative result on a serum or urine pregnancy test within 1 week prior to the procedure.

Willingness to allow storage of blood or biopsy samples for possible future use to study HIV/AIDS, related diseases or the immune system; willingness to permit HLA testing.

FOR PATIENTS UNDERGOING BIOPSIES:

No medical contraindication to tonsillar, lymph node, or intestinal biopsy.

For tonsillar biopsy, presence of visible tonsillar tissue; for lymph node biopsy, palpable lymph nodes.

No aspirin or piroxicam (Feldene) for 10 days prior to the procedure; other non steroidal anti-inflammatory drugs (e.g. ibuprofen) must be discontinued the day prior to the procedure. Acetaminophen [Tylenol] is permitted at any time.

FOR PATIENTS UNDERGOING BAL:

Hematocrit greater than 27 percent, platelets greater than 50,000/ml.

Baseline pulse-oximetry recording of 94 percent or greater unless clinical indication for bronchoscopy.

No medical contraindication to bronchoscopy.

In addition to the above:

FOR HIV POSITIVE VOLUNTEERS:

HIV infection must be confirmed by ELISA and western blot or dot blot. For patients with acute HIV infection and negative HIV serology, plasma HIV viral load greater than 10,000 copies/ml.

FOR HEALTHY VOLUNTEERS:

No underlying significant medical problem, especially an immunodeficiency or autoimmune disease, or an underlying problem requiring immunosuppressive therapy.

Absence of HIV infection as confirmed by negative ELISA and, if indicated, western blot or dot blot.

FOR ICL PATIENTS:

Patients must meet the definition of ICL according to the CDC criteria: documented absolute CD4 T lymphocyte count of less than 300 cells per cubic millimeter or of less than 20 percent of total T cells on more than one occasion usually two to three months apart, without evidence of HIV infection or any defined immunodeficiency or therapy associated with depressed levels of CD4 T cells.

Absence of HIV infection as confirmed by negative ELISA and, if indicated, western blot or dot blot.

EXCLUSION CRITERIA:

FOR ALL VOLUNTEERS UNDERGOING BIOPSIES:

Platelet count less than 75,000 platelets/mm(3).

PT or PTT prolonged by greater than 2 seconds unless patient has documented lupus anticoagulant/anti-phospholipid syndrome, which is not associated with an increased bleeding risk

Known underlying bleeding disorder.

Pregnancy.

FOR HIV-POSITIVE OR ICL VOLUNTEERS FOR LYMPH NODE BIOPSIES:

Use of narcotics (other than as prescribed by a physician) or cocaine less than 1 week prior to the date of biopsy.

FOR ALL VOLUNTEERS FOR INTESTINAL BIOPSIES:

Use of narcotics (other than as prescribed by a physician) or cocaine less than 1 week prior to the date of biopsy.

Significant heart valve abnormalities.

Presence of pacemaker, artificial joint or vascular surgery graft.

FOR ALL VOLUNTEERS FOR BAL:

Use of narcotics (other than as prescribed by a physician) or cocaine less than 1 week prior to the date of biopsy.

Pregnancy.

Any medical condition for which the investigators believe bronchoscopy may be contraindicated.

Allergy to lidocaine.

History of asthma requiring therapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include patients already seen in our outpatient clinic, as well as individuals recruited from outside clinics.
Sampling Method: Non-Probability Sample
Enrollment: 635 (Estimated)
Dates: Start 1994-11-30 (Actual)

PRIMARY OUTCOMES:
Obtain lymphoid tissue by tonsillar, lymph node, or intestinal biopsies, or BAL fluid in patients with HIV, ICL, and healthy volunteers to evaluate for viral burden, lymphocyte subsets, and cytokine production. | Each procedure visit where tissue is obtained.
  Evaluate for viral burden, lymphocyte subsets, and cytokine production.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Zeng M, Southern PJ, Reilly CS, Beilman GJ, Chipman JG, Schacker TW, Haase AT. Lymphoid tissue damage in HIV-1 infection depletes naive T cells and limits T cell reconstitution after antiretroviral therapy. PLoS Pathog. 2012 Jan;8(1):e1002437. doi: 10.1371/journal.ppat.1002437. Epub 2012 Jan 5. PMID 22241988
- [Background] Brenchley JM, Schacker TW, Ruff LE, Price DA, Taylor JH, Beilman GJ, Nguyen PL, Khoruts A, Larson M, Haase AT, Douek DC. CD4+ T cell depletion during all stages of HIV disease occurs predominantly in the gastrointestinal tract. J Exp Med. 2004 Sep 20;200(6):749-59. doi: 10.1084/jem.20040874. Epub 2004 Sep 13. PMID 15365096
- [Background] Mavigner M, Cazabat M, Dubois M, L'Faqihi FE, Requena M, Pasquier C, Klopp P, Amar J, Alric L, Barange K, Vinel JP, Marchou B, Massip P, Izopet J, Delobel P. Altered CD4+ T cell homing to the gut impairs mucosal immune reconstitution in treated HIV-infected individuals. J Clin Invest. 2012 Jan;122(1):62-9. doi: 10.1172/JCI59011. Epub 2011 Dec 12. PMID 22156200
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1995-I-0027.html